CLINICAL TRIAL: NCT01684683
Title: Clinical Efficacy and Safety of Theophylline in the Treatment of Non-Cystic Fibrosis(NCF) Bronchiectasis
Brief Title: The Effect of Theophylline in the Treatment of Bronchiectasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Xugang, Doctor of Medicine, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: theophylline in NCFB
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Theophylline; Therapeutic Uses; HDAC; HAT; Random placebo study
MeSH Terms: conditions — Bronchiectasis | interventions — Theophylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Theophylline (Experimental): Theophylline sustained-release tablet by mouth 100mg every 12hours for 24weeks
  Interventions: Drug: Theophylline
- placebo (Placebo Comparator): Placebo(for Theophylline sustained-release tablet) tablet by mouth 100mg every 12hours for 24weeks
  Interventions: Drug: Placebo(for Theophylline)

INTERVENTIONS:
Drug: Theophylline — Theophylline 0.1 bid
  Other Names: Theophylline Sustained-Release Tablet.
  Arms: Theophylline
Drug: Placebo(for Theophylline) — Starch tablet manufactured to Theophylline 100mg (Theophylline Stained-Release Tablet)
  Arms: placebo

SUMMARY:
Theophylline was well recommended in the treatment of chronic obstructive pulmonary disease (COPD) and asthma. However, there is no supporting evidence for their efficacy in the treatment of bronchiectasis. Our hypothesis is that theophylline will play a role in bronchiectasis. Our purpose is to examine the efficacy and safety of 24 weeks treatment with theophylline in subjects with non-cystic fibrosis bronchiectasis.

DETAILED DESCRIPTION:
For the reasons of lack of sufficient clinical trial evidences, there are no standard therapy recommendations for bronchiectasis. Currently the treatments for bronchiectasis are mostly based on experience gained from the treatment of COPD and cystic fibrosis(CF). The aims of treatment for bronchiectasis are to improve the health-related quality of life, to slow down the decrease of lung function, to reduce the exacerbation frequence and the mortality. The mechanism of treatment are including: treating the underlying disease; improving drainage of sputum; anti-infection; anti-inflammation; treating airway obstruction. A review written by Peter J. Barnes describes that as a bronchodilator in COPD, theophylline may relax human airways smooth muscle, have an anti-inflammation rols, and have an additional effect on mucociliary clearance. Besides, theophylline can improve the activity of histone deacetylase, which will reverse the resistant of corticosteroids. We hypothesis that theophylline will have the same effect in subjects with NCF-bronchiectasis as in subjects with COPD. Our trial may give an evidence of using theophylline in treatment of bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-70 years old with non-CF bronchiectasis ,free from acute exacerbations for at least 3 months.Stable phase of the disease.

Exclusion Criteria:

* Patients with a cigarette smoking history of more than 10 packs-year. Patients with COPD. Patients with traction bronchiectasis due to advanced fibrosis. Patients with known intolerance for theophylline. Patients with asthma. Patients with other disease disturbing outcomes of the trials. Patients without consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Scores of the St.George's Respiratory Questionnaire | At 24 weeks

SECONDARY OUTCOMES:
The Number of Exacerbations | At 24 weeks
Scores of The Leicester Cough Questionnaire | At 24 weeks
24 Hour Sputum Volume | Every day for 24 weeks
Activity of histone deacetylase(HDAC) | At 24 weeks
  HDACs are extracted from cells in blood.
Activity of histone acetyltransferase(HAT) | At 24 weeks
  HATs are extracted from cells in blood.
Lung function | At 24 weeks
  Lung function as measured by FEV1, FVC, FEV1%, FEV1/FVC, FEF25-75 values following American Thoracic Society(ATS) guidelines
Induced sputum culture | At 24 weeks
Induced Sputum Cytology Count | At 24 weeks
Interleukin-6(IL-6) | At 24 weeks
  Test IL-6 both in blood and sputum.
C-Reactive Protein | At 24 weeks
To evaluate change in patients' Clinical Data | Every day for 24 weeks
  Clinical Data contain dyspnea, cough, wheezes, hemoptysis, sputum characteristics, sputum volume.
Number of participants with adverse events | Up to 24 weeks
  Adverse events may contain symptoms such as nausea, sickness, headache, insomnia, palpitation, arrhythmia and so on. Record the symptoms and times of the patients.
Plasma Concentration of Theophylline | At 24 weeks
  Venous blood was taken for plasma theophylline at the end of the treatment period. (At the very time of 2 hours after patients taken the pills)
IL-8 | At 24 weeks
  Test IL-8 both in blood and sputum.
IL-10 | At 24 weeks
  Test IL-10 both in blood and sputum.
Human Tumor Necrosis Factor α（TNF-α) | At 24 weeks
  Test TNF-α both in blood and sputum.
8-Isoprostane | At 24 weeks
Blood routine examination | At 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chen Rongchang, Professor, Study Director — institute vice director; Zhong Nanshan, Professor, Study Director — institute director
Locations (1):
- State Key Laboratory of Respiratory Research Institute., Guangzhou, Guangdong, China